CLINICAL TRIAL: NCT02887222
Title: Programmed Intermittent Epidural Bolus for Labor Analgesia During First Stage of Labor: A Sequential Allocation Trial to Determine the Optimum Interval Time Between Boluses of a Fixed Volume of 5 ml of Bupivacaine 0.125% Plus Fentanyl 2 mcg/ml
Brief Title: Programmed Intermittent Epidural Bolus for Labor Analgesia During First Stage of Labor-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-06
Record Dates: First submitted 2016-08-29; First posted 2016-09-02 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Labor Pain
Keywords: Epidural; Labor analgesia; Programmed intermittent epidural bolus
MeSH Terms: conditions — Labor Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- PIEB volume of 7 mL (Active Comparator): The infusion pump will deliver programmed intermittent epidural boluses at a 40-minute interval. The bolus will consist of 7mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml. A PCEA bolus of 5mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml will also be available.
  Interventions: Drug: Bupivacaine
- PIEB volume of 8 mL (Active Comparator): The infusion pump will deliver programmed intermittent epidural boluses at a 40-minute interval. The bolus will consist of 8mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml. A PCEA bolus of 5mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml will also be available.
  Interventions: Drug: Bupivacaine
- PIEB volume of 9 mL (Active Comparator): The infusion pump will deliver programmed intermittent epidural boluses at a 40-minute interval. The bolus will consist of 9mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml. A PCEA bolus of 5mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml will also be available.
  Interventions: Drug: Bupivacaine
- PIEB volume of 10 mL (Active Comparator): The infusion pump will deliver programmed intermittent epidural boluses at a 40-minute interval. The bolus will consist of 10mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml. A PCEA bolus of 5mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml will also be available.
  Interventions: Drug: Bupivacaine
- PIEB volume of 11 mL (Active Comparator): The infusion pump will deliver programmed intermittent epidural boluses at a 40-minute interval. The bolus will consist of 11mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml. A PCEA bolus of 5mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml will also be available.
  Interventions: Drug: Bupivacaine
- PIEB volume of 12 mL (Active Comparator): The infusion pump will deliver programmed intermittent epidural boluses at a 40-minute interval. The bolus will consist of 12mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml. A PCEA bolus of 5mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml will also be available.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — 0.0625% Bupivacaine plus fentanyl 2mcg/ml
  Other Names: Marcaine

SUMMARY:
Until recently, at Mount Sinai Hospital (MSH), epidural analgesia for labor pain was delivered with a pump that could only provide continuous infusion of the freezing medication in combination of pushes of medication activated by the patient, a technique called patient controlled epidural analgesia (PCEA). In the last decade or so, the literature has suggested that this continuous infusion of medication is not as effective as previously thought, and suggested that instead of continuous infusion we should use intermittent programmed pushes. The investigators now have devices that are able to do that. Programmed intermittent epidural bolus (PIEB) is a new technological advance based on the concept that boluses of freezing medication in the epidural space are superior to continuous epidural infusion (CEI). Recently the epidural pumps at MSH were reprogrammed to deliver bolus of medication at regular intervals (PIEB), in addition to what the patient can deliver herself (PCEA). Studies have shown that delivering analgesia in this manner prolong the duration of analgesia, reduce motor block, lower the incidence of breakthrough pain, improve maternal satisfaction and decrease local anesthetic consumption. The investigators have recently concluded a study at MSH using PIEB where excellent results were observed. However, in that study, some patients exhibited higher than necessary sensory blocks. The investigators believe that the technique can be optimized by using the same interval of the previous study with smaller volumes of the intermittent boluses. Optimizing the technique, may allow the investigators to be able to reduce even further the amount of medication used by each patient.

The hypothesis of this study is that there is an optimal volume of the PIEB bolus at a fixed interval of 40 minutes of 0.0625% bupivacaine plus fentanyl 2mcg/ml that will provide 90% of women the necessary drug requirements during first stage of labor (EV90), thus avoiding breakthrough pain and need for PCEA or physician intervention. We hypothesize that this effective volume will be between 7 and 12 mL (6.6 mg/hr to 11.3 mg/hr of bupivacaine).

DETAILED DESCRIPTION:
Studies involving programmed intermittent epidural bolus (PIEB) to date have provided an analgesic regimen that delivered an amount of local anesthetic that was below the patient's requirement per hour, as the studies were done in the context of an association with patient controlled epidural anesthesia (PCEA) as a rescue technique. As a result, PCEA requests were frequent and therefore these studies have not been able to truly understand the pharmacology of the bolus technique in the PIEB regimen, as the PCEA utilized by patients added an extra component to the regimen.

At Mount Sinai Hospital, PIEB devices have been recently introduced. Currently our standard epidural mixture is bupivacaine 0.0625% with fentanyl 2mcg/ml. Based on previous research done by the investigators, the current epidural regimen consists of 10 ml PIEB at 40 minute intervals, with PCEA boluses of 5 ml and a lock out interval of 10 minutes, for a maximum of 20 ml of the epidural mixture per hour.

In this study, the investigators will vary the volume of the bolus (7-12 mL) of bupivacaine 0.0625% with fentanyl 2mcg/ml. PCEA bolus of 5mL of the same solution will also be available. The goal is to establish the ideal PIEB volume that will be effective for our patient population.

ELIGIBILITY:
Inclusion Criteria:

* ASA 2 or 3
* ≥ 37 weeks gestation
* nulliparous
* Singleton pregnancy, vertex presentation
* Active labor: regular painful contractions occurring at at least every 5 minutes and change in cervix
* Verbal Numerical Pain Score (VNPS) at requesting analgesia > 5 (VNPS 0-10)
* Cervical dilatation ≥2 ≤ 5 cm

Exclusion Criteria:

* Refusal to provide written informed consent
* Patients unable to communicate fluently in English
* Any contraindication to epidural anesthesia
* Unintentional dural puncture
* Allergy or hypersensitivity to bupivacaine or fentanyl
* Use of opioids or sedatives within the last 4 hours.

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Adequate response of the patient, defined as no request for supplemental analgesia | 6 hours
  Adequate response of the patient, defined as no request for supplemental analgesia (PCEA bolus or clinician administered bolus) until the completion of the first stage of labor or until 6 hours following initiation of the programmed intermittent epidural bolus (PIEB).

SECONDARY OUTCOMES:
Sensory block level to ice | 6 hours
  Sensory block to ice will be assessed bilaterally at the mid axillary lines, and the level of block will be the level at which the patient still does not feel normal cold sensation as compared to a control site (lateral upper arm).
Sensory block level to pin prick | 6 hours
  Sensory block to pin prick will be assessed bilaterally at the mid axillary lines, and the level of block will be the level at which the patient initial begins to feel normal sharp sensation compared to a control site (lateral upper arm).
Motor block level assessed using Bromage score | 6 hours
  Motor block will be assessed with the Bromage score: 0 = able to raise the extended leg; 1 = unable to raise the extended leg but able to flex knees; 2 = unable to flex knees, but able to flex ankle; 3 = unable to flex ankle.
Hypotension | 6 hours
  A decrease in systolic blood pressure greater than 20% from baseline (defined as an average of 3 readings prior to epidural).
Pain score | 6 hours
  Pain score measured hourly using VNRS (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No